CLINICAL TRIAL: NCT01665495
Title: Drainage or Pericardiocentesis Alone for Recurrent Non-malignant Pericardial Effusions Requiring Intervention.
Brief Title: Drainage or Pericardiocentesis (DROP) Alone for Recurrent Non-malignant Pericardial Effusions Requiring Intervention
Acronym: DROP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maria Vittoria Hospital (Other)
Responsible Party: Principal Investigator, Massimo Imazio, Cardiologist, Maria Vittoria Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 72/16/11
Record Dates: First submitted 2012-08-12; First posted 2012-08-15 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Pericardial Effusion
Keywords: pericardial effusion; cardiac tamponade; pericardiocentesis; pericardial drainage; prevention
MeSH Terms: conditions — Pericardial Effusion; Cardiac Tamponade

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pericardiocentesis (No Intervention): Pericardial fluid drained by simple echo-guided pericardiocentesis
- Extended pericardial drainage (Active Comparator): Extended pericardial drainage will include pericardiocentesis followed by an intermittent pericardial catheter drainage. Pericardial drainage will be kept till daily fluid return<30ml
  Interventions: Procedure: Extended pericardial drainage by catheter

INTERVENTIONS:
Procedure: Extended pericardial drainage by catheter — Extended pericardial drainage will be done after pericardiocentesis by the insertion of a catheter to intermittently drain pericardial fluid till daily fluid return<30 ml.
  Arms: Extended pericardial drainage

SUMMARY:
The DROP study is a prospective, multi center, randomized, open-label trial to test the efficacy and safety of extended catheter pericardial drainage in patients with non-malignant pericardial effusions.

DETAILED DESCRIPTION:
The trial will compared the efficacy and safety of pericardiocentesis alone compared with extended pericardial catheter drainage for the prevention of recurrent effusions in patients with non-malignant pericardial effusions requiring intervention.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* pericardial effusion requiring pericardiocentesis
* non-malignant etiology

Exclusion Criteria:

* known neoplastic etiology
* known bacterial etiology

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Recurrent pericardial effusion | 12 months
Need for repeated pericardiocentesis | 12 months
Need for cardiac surgery | 12 months

SECONDARY OUTCOMES:
Hospital stay | 12 months
Disease-related hospitalization | 12 months
Overall mortality | 12 months

OTHER OUTCOMES:
Complication rates | 12 months
  Major complications: fatal, life-threatening or requiring any intervention Minor complications: any requiring only monitoring or follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Imazio, MD, Principal Investigator — Cardiology Department, Maria Vittoria Hospital
Locations (7):
- Italy (7):
  - Ospedali Riuniti, Bergamo
  - Ospedale Regionale San Maurizio, Bolzano
  - Ospedale Niguarda, Milan
  - Ospedale degli Infermi, Rivoli
  - Cardiology Department, Maria Vittoria Hospital, Torino
  - Cardiology Department, Ospedale San Giovanni Bosco, Torino
  - Ospedale Mauriziano, Torino

REFERENCES:
- [Derived] Imazio M, Belli R, Beqaraj F, Giammaria M, Lestuzzi C, Hoit B, LeWinter M, Spodick DH, Adler Y; DROP Investigators. DRainage Or Pericardiocentesis alone for recurrent nonmalignant, nonbacterial pericardial effusions requiring intervention: rationale and design of the DROP trial, a randomized, open-label, multicenter study. J Cardiovasc Med (Hagerstown). 2014 Jun;15(6):510-4. doi: 10.2459/JCM.0b013e3283621d26. PMID 23867908